CLINICAL TRIAL: NCT05311072
Title: A Chinese Real-world Study to Investigate the Management Pattern and Outcomes of Chronic Thromboembolic Pulmonary Hypertension (CHANGE Study)
Brief Title: Change-a Multi-center Chronic Thromboembolic Pulmonary Hypertension （CTEPH） Database in China
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: Change-CTEPH
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic Thromboembolic Pulmonary Hypertension; epidemiology; diagnosis; treatment; prognosis; balloon pulmonary angioplasty; pulmonary endarterectomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood samples and PEA specimens of patients with CTEPH
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PEA cohort: patients with CTEPH receiving PEA
  Interventions: Procedure: pulmonary endarterectomy or balloon pulmonary angioplasty
- BPA cohort: patients with CTEPH receiving BPA
  Interventions: Procedure: pulmonary endarterectomy or balloon pulmonary angioplasty
- Pulmonary arterial hypertension (PAH)-specific medication: CTEPH patients without PEA or BPA, treatment with any PAH-specific medication, i.e. endothelin receptor antagonists, phosphodiesterase type 5 inhibitors, soluble guanylate cyclase stimulators, drugs acting on the prostanoid pathway and prostaglandin I2 receptor agonists
  Interventions: Procedure: pulmonary endarterectomy or balloon pulmonary angioplasty

INTERVENTIONS:
Procedure: pulmonary endarterectomy or balloon pulmonary angioplasty — A multidisciplinary team make the final treatments for patients with CTEPH depending on their disease and preferences.
  Other Names: PEA or BPA

SUMMARY:
The Change Database is a prospective, observational multi-center disease registry, which will collect data on patients with chronic thromboembolic pulmonary hypertension (CTEPH) in China. It aims to illustrate the epidemiology, management and long-term outcomes of CTEPH.

DETAILED DESCRIPTION:
18 CTEPH centers will be enrolled in the study. The epidemiology, diagnosis，treatments (pulmonary endarterectomy (PEA), balloon pulmonary angioplasty (BPA) and targeted medical therapy), and long-term prognosis of CTEPH will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with chronic thromboembolic pulmonary hypertension (CTEPH)
2. Patients must be willing to provide informed consent
3. Patients must meet the following criteria for CTEPH:

a mean pulmonary artery pressures (mPAP) ≥20 mmHg combined with a pulmonary vascular resistance (PVR) ≥ 3 WU and pulmonary arterial wedge pressure (PAWP)≤ 15 mmHg documented at right heart catheterization with radiographic evidence of organized thrombi involving the pulmonary arteries after 3 months of effective anticoagulation.

Exclusion Criteria:

1. Main cause of PH other than CTEPH
2. Participation in a therapeutic clinical trial with an unknown drug;
3. Withdrawal or lack of informed consent.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients dianosed with CTEPH according to the contemporary guidelines
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
death | 3 years
  all-cause death
The change in mean pulmonary artery pressure (mPAP) in millimetre of mercury (mmHg), pulmonary vascular resistance (PVR) in Wood units, cardiac output (CO) in liter per minute (L/min) or cardiac index (CI) in liter per minute (L/min). | 3 years
  mPAP, PVR, CO, and CI constitute critical parameters in hemodynamic assessments.
The change in 6-minute walk distance in meter, in BNP or NT-proBNP in picograms per milliliter（pg/ml), or WHO-functional class. | 3 years
  The 6-minute walk distance, BNP or NT-proBNP levels, and WHO-functional class are parameters used in the evaluation of functional capacity.

SECONDARY OUTCOMES:
lung or heart and lung transplantation | 3 years
  proportion of patients experiencing lung or heart and lung transplantation due to severe right heart failure during the study
changes of health related quality of life | 3 years
  change of quality of life measured with the EQ-5D-5L or EmPHasis-10

OTHER OUTCOMES:
bleeding | up to 3 years
  fatal bleeding, major bleeding, clinically relevant non-major bleeding, based on the ISTH definition
symptomatic recurrence of DVT or PE | up to 3 years
  reappearance of clinical manifestations or symptoms associated with DVT or PE after a previous episode or treatment, include leg pain, swelling, warmth, redness, or shortness of breath,etc
complication of treatment interventions (PEA or BPA) | up to 3 years
  complications include lung injury, haemoptysis, residual pulmonary hypertension, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Frendship hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Li Y, Yang Y, Gong S, Yang Z, Hong C, Cui X, Wan J, Ji Y, Chen H, Zhu L, Li C, Cheng Z, Zhang Y, Wang Q, Luo Q, Guo L, Ma G, Han B, Liu Z, Xiong C, Wang L, Ji Q, Li F, Wang S, Zhang Z, Zhang Y, Wang D, Gao Q, Huang Q, Xie W, Zhai Z, Wang C. The management pattern and outcomes of chronic thromboembolic pulmonary hypertension: rationale and design for a Chinese real-world study. BMC Pulm Med. 2024 Jun 3;24(1):265. doi: 10.1186/s12890-024-03042-5. PMID 38825688